CLINICAL TRIAL: NCT05641623
Title: OSU6162 as add-on in SSRI/SNRI-resistant Depression (ODEN): a Double-blind, Placebo-controlled Evaluation of Efficacy and Safety
Brief Title: OSU6162 as add-on in SSRI/SNRI-resistant Depression
Acronym: ODEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Arvid Carlsson Research AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT number: 2020-005860-69; 2024-513894-35-00 (EU CTIS Number); 2020-005860-69 (EudraCT Number)
Record Dates: First submitted 2021-11-11; First posted 2022-12-07 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Depression; Depressive Disorder, Treatment-Resistant; Depressive Disorder; Depressive Episode; Recurrent Depressive Disorder; Recurrent Depression
Keywords: Antidepressant; drug therapy, combination; Dopamine Drugs; Dopamine; Selective Serotonin Reuptake Inhibitor; SNRI; SSRI; Serotonin and Norepinephrine Reuptake Inhibitors
MeSH Terms: conditions — Depression; Depressive Disorder, Treatment-Resistant; Depressive Disorder | interventions — OSU 6162; 3-(3-(methylsulfonyl)phenyl)-1-propylpiperidine

STUDY DESIGN:
Intervention Model Description: Double-blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Monitor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSU6162 (Active Comparator): White, circular, coated tablets. Flexible dosage: the starting dose will be 15 mg TID and the maximal dose 45 mg TID.
  Interventions: Drug: OSU6162
- Placebo (Placebo Comparator): Coated tablets, flexible dosage, TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OSU6162 — OSU6162
  Other Names: OSU-6162; PNU-96391
  Arms: OSU6162
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomised, placebo-controlled, parallel-group trial comparing OSU6162 at flexible dosage with placebo as add-on to treatment with an SSRI/SNRI in patients with depression that have not responded to treatment with an SSRI/SNRI per se for at least 6 weeks. The study will last for 6 weeks, after which those not having responded will leave the trial and those having responded will be offered to continue treatment without unblinding for another 4 weeks. Optional Substudy 1 and 2: Baseline and treatment-associated change in reward-related striatal activity per fMRI-assessment. (Substudy 1).

Brain signal variability per fMRI-assessment. (Substudy 1). Probabilistic Reward Task (PRT). (Substudy 2).

While assessment of the efficacy and safety of OSU6162 is the main objective of this study, possible differences between the two treatment groups with respect to a number of biomarkers in serum will also be explored.

Multicenter trial: Multiple sites four Gothenburg, Lund, Stockholm and Uppsala.

DETAILED DESCRIPTION:
The treatment period will be 6 weeks during which all subjects will make 7 study visits and be in contact with study nurse or physician by phone at 4 occasions. The first visit is a screening visit followed by a baseline visit for inclusion and start of treatment with OSU6162 or placebo.

Optional for the subjects Substudy 1 and 2: Baseline and treatment-associated change in reward-related striatal activity per fMRI-assessment. (Substudy 1).

Brain signal variability per fMRI-assessment. (Substudy 1). Probabilistic Reward Task (PRT). (Substudy 2).

Those responding to treatment will be offered to participate in the extension phase of the study for an additional 4 weeks during which the subjects will make 3 study visits and take 3 telephone interviews.

Before inclusion in the study, all subjects will be informed both verbally and in writing about its purpose, its procedures, and possible risks associated with participation. Before any study-specific procedures take place, written informed consent will be obtained.

Multicenter trial. Multiple sites 4: Sahlgrenska University Hospital Gothenburg, Skåne University Hospital Psychiatry Lund, North Stockholm psychiatry Stockholm region and Uppsala University Hospital Department of neuroscience Uppsala.

For participation in the extension phase, four factors must be fulfilled: 1. The subject must regard himself/herself as clearly improved and be willing to continue. 2. The investigator must assess the subject as clearly improved. 3. The subject must display at least 50% reduction on HDRS6 as compared to baseline. 4. The subject must have signed a new informed consent.

While assessment of the efficacy and safety of OSU6162 is the main objective of this study, possible differences between the two treatment groups with respect to a number of biomarkers in serum will also be explored.

The primary evaluation of efficacy will be undertaken at the endpoint of the 6-week trial. All analyses will however be repeated also at the endpoint of the 4-week extension phase for subjects participating in this part of the study.

Data will be analysed using mixed models for repeated measurement which means that the model includes data from all depression ratings from baseline to endpoint; this method, which is usually recommended to be used in depression trials by the authorities, is considered to handle data loss due to patients leaving a study prematurely in a better way than imputation methods such as the last observation carried forward (LOCF) technique.

ELIGIBILITY:
Inclusion Criteria

In order to be included in the study, subjects must meet the following criteria:

1. Signed informed consent.
2. Age: 25-65 on the day of screening.
3. Meeting DSM-5 criteria for major depressive disorder as confirmed by the Mini International Neuropsychiatric Interview (MINI).
4. A symptom-free period preceding the current episode within the past two years confirmed at interview.
5. Not significantly improved, as judged by both doctor and patient, after having been treated with one of the following SSRIs/SNRIs: citalopram, escitalopram, paroxetine, sertraline, fluoxetine, duloxetine, or venlafaxine for at least 6 weeks.
6. Displaying a sum score of MADRS ≥22.
7. In women of childbearing potential (WOCBP): negative result of a pregnancy test and a method of contraception with a failure rate of less than 1 %. Contraception must be used during the treatment and follow-up period. Acceptable forms of contraception are:

   1. Use of combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation

      * oral
      * intravaginal
      * transdermal
   2. progestogen-only hormonal contraception associated with inhibition of ovulation:

      * oral
      * injectable
      * implantable
   3. Placement of intrauterine device (IUD) or intrauterine hormone releasing system (IUS)
   4. Bilateral tubal occlusion or ligation
   5. Vasectomised partner (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate and provided that male partner is the sole sexual partner of the WOCBP trial participant).
   6. Sexual abstinence.
8. Male patients must agree to use condoms during the study and for 2 weeks after the end of the study/last dose of IMP, unless their partner is using a highly efficient method of contraception, as described above.

Exclusion criteria

Subjects must not be included in the study if any of the following criteria are met:

1. Meeting MINI criteria at interview for suicidality, manic episode, hypomanic episode, bipolar I, bipolar II, bipolar unspecified, bipolar I with psychotic symptoms, panic disorder (current), agoraphobia, posttraumatic stress disorder, alcohol dependency, alcohol abuse, substance dependency (non-alcoholic), substance abuse (non-alcoholic), psychotic disorders, mood disorders with psychotic features, anorexia nervosa, bulimia nervosa, anorexia nervosa binge eating / purging type, or antisocial personality disorder.

   Meeting MINI criteria at interview for generalised anxiety disorder, obsessive compulsive disorder or social anxiety (social phobia), unless the present symptoms can predominantly be attributed to a diagnosis of major depressive disorder.
2. A history of substance/alcohol abuse within 2 years prior to screening.
3. A previous diagnosis of a personality disorder, autism spectrum disorder, attention-deficit/hyperactivity disorder, or intellectual disability.
4. Any other previously diagnosed or suspected CNS disorder that according to the investigator renders the patient unsuitable for participation in the trial.
5. Any factor that according to the investigator renders it unlikely that the patient will comply with the instructions regarding treatment, visits etc.
6. Any somatic illness that according to the investigator renders the patient unsuitable for participation in the trial.
7. Any signs or symptoms of somatic illness resulting from assessment of vital signs, physical examination, clinical laboratory tests, and 12-lead ECG that according to the investigator renders the patient unsuitable for participation for safety reasons, including a QTc-time on ECG exceeding 450 ms in men and 460 ms in women.
8. Any change in dosage of said SSRI/SNRI within 4 weeks prior to screening or at any time during the course of the trial.
9. Treatment with any other psychoactive drug than said SSRI/SNRI with the exception of using mirtazapine up to 15 mg for sleep, occasional use of benzodiazepines and benzodiazepine-like anxiolytics or hypnotics and occasional use of antihistaminergic sedatives (without anti-dopaminergic effects) within 4 weeks prior to screening and at any time during the course of the trial.
10. Patients who are receiving concomitant therapy with potent cytochrome P450 enzyme inhibitors (e.g., bupropion, fluvoxamin, ketoconazole, itraconazole, telithromycin, clarithromycin, protease inhibitors, quinidine, and terbinafine).
11. Ongoing treatment with drugs with a narrow therapeutic window where either lower or higher serum levels are potentially harmful (including but not limited to warfarin along with other anticoagulants, digoxin along with other antiarrythmics, anticonvulsants prescribed for treatment of epilepsy, cyclosporine, immunosuppressants, and lithium).
12. Current treatment with any prescribed or OTC drug that according to the investigator renders the subject unsuitable for participation in the trial.
13. Previous intake of OSU6162.
14. Current participation in another clinical trial.
15. Nursing women.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Bech 6-item subscale of the Hamilton Depression Rating Scale (HDRS) | Endpoint at 42 days treatment
  Change from baseline with respect to the total score of the investigator-rated Bech 6-item subscale of the Hamilton Depression Rating Scale (HDRS) at endpoint.
  Lower scores mean a better outcome.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale (HDRS) | Endpoint at 42 days treatment
  Number of participants displaying clinical response defined as ≥50% reduction in the total score of the investigator-rated Bech 6-item subscale of the HDRS.
  Number of participants displaying clinical remission defined as a sum rating of ≤4 in the total score of the investigator-rated Bech 6-item subscale of the HDRS.
  Change from baseline with respect to investigator-rated item 1 (depressed mood) of the HDRS.
  Change from baseline with respect to the total score of the investigator-rated HDRS.
  Lower scores mean a better outcome.
Investigator-rated Montgomery Åsberg Depression Rating Scale (MADRS) | Endpoint at 42 days treatment
  Change from baseline with respect to the total score. Lower scores mean a better outcome.
investigator-rated Clinical Global Impression - Severity scale (CGI-S) | Endpoint at 42 days treatment
  Change from baseline with respect to the total score. Lower scores mean a better outcome.
Clinical Global Impression - Change scale (CGI-C) | Endpoint at 42 days treatment
  Investigator rating. Lower scores mean a better outcome.
Patient-rated Fatigue Severity Scale (FSS) | Endpoint at 42 days treatment
  Change from baseline with respect to the total score. Lower scores mean a better outcome.
Patient-rated MADRS-S (self) | Endpoint at 42 days treatment
  Change from baseline with respect to the total score. Lower scores mean a better outcome.
Patient-rated Snaith-Hamilton Pleasure Scale (SHAPS) | Endpoint at 42 days treatment
  Change from baseline with respect to the total score. Lower scores mean a better outcome.
Global Rating of Change Scale (GRC) | Endpoint at 42 days treatment
  Patient rating. Lower scores mean a better outcome.
Bech 6-item subscale of the HDRS | Endpoint at 42 days treatment
  Change from baseline with respect to the total score of the investigator-rated Bech 6-item subscale of the HDRS at endpoint in patients displaying a sum rating of ≥36 at the Fatigue Severity Scale at baseline.
  Lower scores mean a better outcome.
Patient Global Rating of Change Scale (GRC) | Endpoint at 42 days treatment
  Patient rating of the Global Rating of Change Scale (GRC) at endpoint in patients displaying a sum rating of ≥36 at the Fatigue Severity Scale at baseline.
  Lower scores mean a better outcome.
Possible markers of depression | Endpoint at 42 days treatment
  Change from baseline to endpoint with respect to serum levels of a number of possible markers of depression: C-reactive protein (CRP), tumor necrosis factor alpha (TNFα), brain-derived neurotrophic factor (BDNF) and interleukin-6 (IL-6).
AE/SAE | Through study completion
  Number of participants with individual AEs and individual SAEs throughout the trial.
Serum levels of medications | Endpoint at 42 days treatment
  Serum levels of OSU6162 at endpoint and of the prescribed SSRI/SNRI at screening and endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Eriksson, Professor, Study Director — Göteborg University
Locations (4):
- Sweden (4):
  - Skåne University Hospital Psychiatry Lund, Lund, Skåne County
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - North Stockholm psychiatry Stockholm region, Stockholm
  - Uppsala University Hospital Department of neuroscience, Uppsala

IPD SHARING:
Plan to Share IPD: No